CLINICAL TRIAL: NCT05051189
Title: Effect of Opioids on Central Control of Ventilation in Children With Obstructive Sleep Apnea
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Houston (Other); Children's Hospital of Philadelphia (Other); Wake Forest University (Other)
Responsible Party: Principal Investigator, Adam Adler MD, MS, FAAP, Associate Professor of Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H50267
Record Dates: First submitted 2021-09-02; First posted 2021-09-21 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: OSA; Opioid; Adenotonsillectomy
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: 2 groups will be identified-
  1. patients with sleep study O2 nadir >85%
  2. patients with sleep study O2 nadir <85%
Who Masked: Participant
Masking Description: The participant will be unaware of the arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patients with sleep apnea having oxygen Saturation >85% randomized to fentanyl 1.0/kg (Active Comparator): Children with OSA having procedures requiring endotracheal intubation and a who will receive opioids (1.0 mcg/kg fentanyl for IBW, max 25 mcg) for evaluation of respiratory changes.
  Interventions: Drug: Fentanyl Citrate
- Patients with sleep apnea having oxygen Saturation <85% randomized to 1.0 mcg/kg fentanyl (Active Comparator): Children without OSA having procedures requiring endotracheal intubation and an who will receive opioids (1.0 mcg/kg fentanyl for IBW, max 25 mcg) for evaluation of respiratory changes
  Interventions: Drug: Fentanyl Citrate
- Patients with sleep apnea having oxygen Saturation >85% randomized to fentanyl 1.5/kg (Active Comparator): Children with OSA having procedures requiring endotracheal intubation and a who will receive opioids (1.5 mcg/kg fentanyl for IBW, max 25 mcg) for evaluation of respiratory changes.
  Interventions: Drug: Fentanyl Citrate
- Patients with sleep apnea having oxygen Saturation <85% randomized to 1.5 mcg/kg fentanyl (Active Comparator): Children with OSA having procedures requiring endotracheal intubation and a who will receive opioids (1.5 mcg/kg fentanyl for IBW, max 25 mcg) for evaluation of respiratory changes.
  Interventions: Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Fentanyl Citrate — Ventilatory response to fentanyl in patients with OSA Specifically: respiratory changes, CO2, RR, TV

SUMMARY:
Children OSA exhibit varying responses to opioids. It is unknown if the degree of intermittent hypoxemia results in different opioid sensitivity

DETAILED DESCRIPTION:
Ventilatory suppression in children following opioid administration is of obvious concern, especially following routine surgical procedures (i.e. adenotonsillectomy). It is thought that patients with obstructive sleep apnea (OSA) have increased sensitivity to opioids, and especially in opioid naïve patients. Recent evidence in children suggests that patients with moderate to severe OSA may not predispose patients to increased opioid sensitivity in the form of respiratory depression when compared with patients that do not have OSA. However, what is not known is wether the degree of hypoxemia experienced by patients effects the opioid sensitivity. The aim of this study is to identify if children with known OSA experience a difference in opioid induced respiratory depression based on the degree of hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing tonsillectomy or adenotonsillectomy
* Ages 2 to up to 8 years
* Preoperative sleep study demonstrating obstructive sleep apnea
* Intubation without medication (e.g. no propofol prior to intubation)
* Requirement for airway instrumentation: LMA or ETT
* Inhalation induction of anesthesia

Exclusion Criteria:

* No obstructive sleep apnea
* Central sleep apnea events >5/hour
* IV induction of anesthesia
* Syndromic patients
* Known or suspected difficult airway
* Allergy to Fentanyl
* Known cardiovascular medications
* Pulmonary hypertension
* Total intravenous anesthesia required
* Parental refusal

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Respiratory depression following opioids | respiratory rate measured at each minute for 10 consecutive minutes following opioid administration
  Identification of respiratory depression following fentanyl administration by recording the respiratory rate prior to and 10 minutes following fentanyl administration
Respiratory depression following opioids | tidal volume measured at each minute for 10 consecutive minutes following opioid administration
  Identification of respiratory depression following fentanyl administration by recording the tidal volume prior to and 10 minutes following fentanyl administration
Respiratory depression following opioids | end tidal co2 measured at each minute for 10 consecutive minutes following opioid administration
  Identification of respiratory depression following fentanyl administration by recording the end-tidal co2 prior to and 10 minutes following fentanyl administration

CONTACTS AND LOCATIONS:
Locations (1):
- Texas childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available at the conclusion of the study upon reasonable written request to the PI
Supporting Information: Study Protocol, SAP, CSR
Time Frame: De-identified raw data will be available upon study completion following written request to the PI. There will be no time restriction on data
Access Criteria: Written request

REFERENCES:
- [Background] Adler AC, Chandrakantan A, Nathanson BH, von Ungern-Sternberg BS. An assessment of opioids on respiratory depression in children with and without obstructive sleep apnea. Paediatr Anaesth. 2021 Sep;31(9):977-984. doi: 10.1111/pan.14228. Epub 2021 Jun 16. PMID 34053151
- [Derived] Adler AC, Lin EE, Messner AH, Rosenberg TL, Pecorella S, Keleghan A, Faircloth S, Templeton TW, Harris L, Khan SA, Pednekar GS, Nguyen DT, Chandrakantan A, von Ungern-Sternberg BS. Association of preoperative nocturnal hypoxaemia nadir and fentanyl ventilatory sensitivity in children with obstructive sleep apnoea undergoing general anaesthesia: a multicentre clinical cohort study. Br J Anaesth. 2025 Nov;135(5):1518-1527. doi: 10.1016/j.bja.2025.07.059. Epub 2025 Sep 5. PMID 40914728